CLINICAL TRIAL: NCT04183244
Title: Efficacy of Erector Spinae Plane Block Versus Infraclavicular Subomohyoid Block in Shoulder Surgery: A Randomized Controlled Blinded Study
Brief Title: Efficacy of Erector Spinae Plane Block Versus Infraclavicular Subomohyoid Block in Shoulder Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Randa Ali Shoukry, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R 57/2019
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain; Shoulder Pain
Keywords: Erector Spinae Plane Block; Infraclavicular Subomohyoid Block; Shoulder Surgery
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae block (Active Comparator): Ultrasound guidance will be used to visualize the transverse processes of T2 and the overlying muscles.
  Under sterile conditions, a 5-cm, 21-gauge needle will be inserted using the out-of-plane technique parallel to the sagittal plane directly over the transverse process,then 30mL of the local anesthetic solution will be injected and observed for the linear spread of LA the under direct ultrasound visualization
  Interventions: Procedure: Erector spinae block
- infraclavicular subomohyoid block (Active Comparator): Performing posterior approach infraclavicular BP block followed by subomohioid block via the same puncture site under ultrasound guidance.
  Interventions: Procedure: Infraclavicular subomohyoid (ISO) block

INTERVENTIONS:
Procedure: Erector spinae block — A 5-cm needle prick in the back of the patient 3 cm lateral to mid-line under sterile conditions, with ultrasound guidance.
  Arms: Erector spinae block
Procedure: Infraclavicular subomohyoid (ISO) block — Under complete aseptic precaution, 12 cm needle will be inserted 2cm superior to the clavicle and advanced retroclavicular, with ultrasound guidance.
  Arms: infraclavicular subomohyoid block

SUMMARY:
The study aimed to compare Erector Spinae Plane (ESP) block versus infraclavicular subomohyoid (ISO) block in the provision of efficacy of either technique in postoperative analgesia in shoulder surgery, aiming to testing the safety of each block in terms of incidence of complications. Patients will be randomly divided into two groups, Group E will receive Erector spinae block and group I will receive infraclavicular subomohyioid block. The local anesthetic solution that will be used in both blocks will be a total volume of 30 mls 0.25%bupivacaine plus 3mg preservative free Dexamethasone. The time between recovery from anesthesia and first pain experienced, as verified by NRS ≥ 3 and first need of a rescue analgesic, will be defined as the duration of analgesia. The total dose of intravenous morphine (the rescue analgesic) used over 24 h postoperatively will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, above 18 years old.
* ASA physical status I
* Scheduled for shoulder surgery

Exclusion Criteria:

* Morbid obese.
* Previous surgery in the same shoulder.
* History of psychiatric disorder.
* Pulmonary disease.
* Contraindication to regional nerve block (e.g. skin infection at the puncture site, coagulopathy).
* Allergy to any of medications that will be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
The block efficacy | 24 hours
  Percentage of 24 hours pain free patients

SECONDARY OUTCOMES:
The incidence of expected complications ( Block safety) | 24 hours
  The incidence of expected complications such as phrenic nerve palsy or pneumothorax.

CONTACTS AND LOCATIONS:
Locations (1):
- Randa Ali Shoukry, Cairo, Al-Nozha, Egypt

IPD SHARING:
Plan to Share IPD: No